CLINICAL TRIAL: NCT01895010
Title: Acupoint Electric Stimulation Combined With Tropisetron in Preventing and Treating Nausea and Vomiting After TACE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, zhu xiao yan, Attending doctor, Fudan University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: ESA2013
Record Dates: First submitted 2013-06-21; First posted 2013-07-10 (Estimated); Last update posted 2013-07-10 (Estimated); Status verified 2013-07

CONDITIONS: Nausea; Vomiting; Metastatic Liver Cancer
Keywords: prevention and treatment; improvement of the patient's appetite; TACE
MeSH Terms: conditions — Nausea; Vomiting; Liver Neoplasms | interventions — Tropisetron

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Acupoint and tropisetron (Experimental): acupoint electric stimulation combined with tropisetron 6mg before TACE
  Interventions: Device: acupoint electric stimulation
- tropisetron (Active Comparator): treated with tropisetron 6mg before TACE
  Interventions: Drug: tropisetron

INTERVENTIONS:
Device: acupoint electric stimulation — acupoint electric stimulation combined with tropisetron 6mg before TACE
  Arms: Acupoint and tropisetron
Drug: tropisetron — only tropisetron 6mg before TACE
  Arms: tropisetron

SUMMARY:
Observation on acupoint electric stimulation combined with tropisetron in preventing and treating nausea and vomiting and improving the patient's appetite after TACE for primary or metastatic liver cancer patients.

DETAILED DESCRIPTION:
* Classification of nausea and vomiting, as measured by NCI CTC-AE version 3
* The improvement of appetite, as measure by the classification of Appetite in accordance with NCI CTC-AE version 3.
* Quality of life: use M. D. Anderson symptom scale (the m. d. Anderson Symptom Inventory,MDASI)

ELIGIBILITY:
Inclusion Criteria:

* ECOG physical status 0,1,2
* would accept the transcatheter hepatic arterial chemoembolization of primary or metastatic liver cancer patients;
* Adult male and female 3, age 18 years old;
* the chem-scheme of arterial infusion chemotherapy based on oxaliplatin dosage of 200mg;
* signed the informed consent and understand the study design;
* Organ function examination in patients must meet the following laboratory indexes: Neutrophil>500/Ul, hemoglobin > 8 gm/dL, platelet >100000/uL,Creatinine < 2 mg/dL bilirubin < 1.5 mg/dL, , alanine aminotransferase < 3 times the normal value, albumin >30g/L
* understand and complete quality of life scale ;
* women of childbearing age urine pregnancy test was negative.

Exclusion Criteria:

* The combined use of other venous chemotherapy within 5 days after TACE;
* skin infection on or near the points;
* skin hyperalgesia, unable to withstand electrical stimulation;
* other confounding factors may cause nausea and vomiting (such as intestinal obstruction, anorexia, etc.);
* heart, cerebrovascular accident history or the history of spinal cord injury;
* intestinal obstruction lead to nausea and vomiting
* installing pacemaker;
* cognitive dysfunction, unable to finish Scale;
* currently using acupuncture therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2013-06; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Classification of nausea and vomiting | 12 month

SECONDARY OUTCOMES:
The improvement of appetite | 12 month

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoyan Zhu, Doc, Principal Investigator — Shanghai Cancer Centre, Fudan University
Locations (1):
- Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Xie J, Chen LH, Ning ZY, Zhang CY, Chen H, Chen Z, Meng ZQ, Zhu XY. Effect of transcutaneous electrical acupoint stimulation combined with palonosetron on chemotherapy-induced nausea and vomiting: a single-blind, randomized, controlled trial. Chin J Cancer. 2017 Jan 10;36(1):6. doi: 10.1186/s40880-016-0176-1. PMID 28069044